CLINICAL TRIAL: NCT02920866
Title: Improving Rehabilitation Outcomes After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: O2251-I; 16-0956 (Other: COMIRB)
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Results first posted 2024-04-29 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty; Osteoarthritis
Keywords: Functional strength integration; Rehabilitation; Hip arthroplasty; Physical function; Muscle performance; Movement compensations
MeSH Terms: conditions — Osteoarthritis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional Strength Integration (FSI) (Experimental): Progressive strength training exercise, specific functional activity to improve pelvic stability and core muscle strength
  Interventions: Behavioral: Functional Strength Integration (FSI)
- Control Group (CON) (Active Comparator): Usual care, continuing education on postsurgical precautions
  Interventions: Behavioral: Control Group (CON)

INTERVENTIONS:
Behavioral: Functional Strength Integration (FSI) — FSI intervention involves strengthening of the hip musculature combined with focused techniques emphasizing early initiation of hip muscle recruitment to stabilize the pelvis, integrating strength and movement pattern training to maximize functional recovery. The FSI program consists of therapeutic exercise in 3 domains: pelvic stability (PST) training, functional training (FT), and strength training (ST). PST includes early surgical-limb weight bearing and core muscle strengthening, progressively increasing in difficulty based on performance benchmarks and therapist monitoring. FT focuses on gait and stair climb exercise, progressing to higher level agility training. ST includes progressive, resistance exercise to improve lower extremity muscle strength. The ST exercises include use of weighted pulleys/weight-training machines. Therapists will determine an 8-rep max for muscle groups and weight will be increased by 10% every 2 weeks to maximize hypertrophy and strength gains.
  Arms: Functional Strength Integration (FSI)
Behavioral: Control Group (CON) — Observed practice patterns from previous investigations and discussion with physical therapists indicate that patients receive rehabilitation services during the 2-3 day hospital stay after THA, but not routinely after hospital discharge. Yet, to control for attention and volume of rehabilitation for the FSI group, patients in the control group will attend outpatient physical therapy for 14 visits (40 minute sessions) over 8 weeks. This control program will mimic the typical postoperative experience for patients in our community, in which patients independently manage their activity. This program will focus on patient education, functional ADL training, and therapeutic exercise. However, the activities in the exercise domain will be limited to low load exercise such as isometric muscle exercise, range of motion (ROM), and flexibility activities. These activities are specifically designed to mirror usual care activity.
  Arms: Control Group (CON)

SUMMARY:
This study plans to learn more about the effects of physical therapy (PT) following a total hip arthroplasty (THA). The purpose of this study is to compare standard of care PT after THA with a physical therapy program specifically designed to integrate targeted core and hip muscle strength and functional training.

DETAILED DESCRIPTION:
Over the next 20 years, the number of total hip arthroplasties (THAs) performed to alleviate pain and disability associated with osteoarthritis (OA) is expected to double to more than 500,000/year. Most patients report improved health-related quality of life following surgery; however, deficits in physical function and quality of life persist. Specifically, Veterans with THA have a higher prevalence of severe activities of daily living (ADL) limitations and report severe physical health-related quality of life deficits. The increased THA utilization, combined with long-term functional deficits which increase heath care utilization, suggests a need for targeted rehabilitation strategies to improve physical function for Veterans after THA.

Movement compensations are a biomarker of functional decline in a variety of older adult populations. For patients with THA, persistent movement compensations are seen in activities of daily living, such as level walking, sit-to-stand transitions, and stair climbing. These movement compensations likely stem from a combination of poor muscle strength and a failure to integrate available muscle strength into functional movement. Functional strength integration (FSI) during daily tasks refers to the ability of the body to produce stable, coordinated movements. At the hip joint, optimal FSI is largely dependent on the ability of hip abductor muscles to produce sufficient hip abduction moments to stabilize the pelvis during unilateral stance tasks. Thus, inability to integrate hip abductor muscle strength during functional tasks results in poor pelvic stability and movement compensations. Lack of FSI possibly explains the deficits in functional recovery after THA. However, current rehabilitation practices do not target the integration of strength and functional movement to resolve movement compensations.

Rehabilitation emphasizing functional strength integration after THA has the potential to substantially improve postoperative physical function by remediating movement compensations with greater hip abductor strength and recruitment during function, providing greater pelvic control and better movement quality. Therefore, the investigators propose a randomized controlled trial of 100 participants to determine if an 8-week functional strength integration (FSI) program after THA improves physical function and muscle performance more than control intervention (CON) after unilateral THA. The secondary goal is to determine if FSI improves movement compensations during functional activity (walking and stair climbing). Eight weeks of intervention will be initiated 2 weeks after THA to allow for early tissue healing. Outcomes will be assessed pre-operatively (PRE); intervention mid-point (after 4 weeks intervention; POST1); intervention end-point (after 8 weeks intervention; POST2) (primary endpoint); and late recovery (26 weeks after initiating rehabilitation; POST3).

ELIGIBILITY:
Inclusion Criteria:

* BMI less than or equal to 40
* Receiving unilateral primary total hip arthroplasty for osteoarthritis

Exclusion Criteria:

* Severe contralateral leg OA (>= 5/10 pain with stair climbing)
* Other unstable orthopaedic conditions that limit function
* Neurological or pulmonary problems that severely limit function
* Uncontrolled hypertension or diabetes
* Use of illegal substances

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sicard-Rosenbaum L, Light KE, Behrman AL. Gait, lower extremity strength, and self-assessed mobility after hip arthroplasty. J Gerontol A Biol Sci Med Sci. 2002 Jan;57(1):M47-51. doi: 10.1093/gerona/57.1.m47. PMID 11773212
- [Result] Jones CA, Voaklander DC, Johnston DW, Suarez-Almazor ME. Health related quality of life outcomes after total hip and knee arthroplasties in a community based population. J Rheumatol. 2000 Jul;27(7):1745-52. PMID 10914862
- [Result] Nilsdotter AK, Isaksson F. Patient relevant outcome 7 years after total hip replacement for OA - a prospective study. BMC Musculoskelet Disord. 2010 Mar 11;11:47. doi: 10.1186/1471-2474-11-47. PMID 20222962
- [Result] Rat AC, Guillemin F, Osnowycz G, Delagoutte JP, Cuny C, Mainard D, Baumann C. Total hip or knee replacement for osteoarthritis: mid- and long-term quality of life. Arthritis Care Res (Hoboken). 2010 Jan 15;62(1):54-62. doi: 10.1002/acr.20014. PMID 20191491
- [Result] Singh JA, Sloan JA. Health-related quality of life in veterans with prevalent total knee arthroplasty and total hip arthroplasty. Rheumatology (Oxford). 2008 Dec;47(12):1826-31. doi: 10.1093/rheumatology/ken381. Epub 2008 Oct 16. PMID 18927190
- [Result] Clough-Gorr KM, Erpen T, Gillmann G, von Renteln-Kruse W, Iliffe S, Beck JC, Stuck AE. Preclinical disability as a risk factor for falls in community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2008 Mar;63(3):314-20. doi: 10.1093/gerona/63.3.314. PMID 18375881
- [Result] Higgins TJ, Janelle CM, Manini TM. Diving below the surface of progressive disability: considering compensatory strategies as evidence of sub-clinical disability. J Gerontol B Psychol Sci Soc Sci. 2014 Mar;69(2):263-74. doi: 10.1093/geronb/gbt110. Epub 2013 Oct 29. PMID 24170713
- [Result] Lamontagne M, Beaulieu ML, Beaule PE. Comparison of joint mechanics of both lower limbs of THA patients with healthy participants during stair ascent and descent. J Orthop Res. 2011 Mar;29(3):305-11. doi: 10.1002/jor.21248. Epub 2010 Sep 30. PMID 20886649
- [Result] Perron M, Malouin F, Moffet H, McFadyen BJ. Three-dimensional gait analysis in women with a total hip arthroplasty. Clin Biomech (Bristol). 2000 Aug;15(7):504-15. doi: 10.1016/s0268-0033(00)00002-4. PMID 10831810
- [Result] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Result] Grimaldi A. Assessing lateral stability of the hip and pelvis. Man Ther. 2011 Feb;16(1):26-32. doi: 10.1016/j.math.2010.08.005. PMID 20888285
- [Result] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Derived] Judd DL, Cheuy VA, Forster JE, Christiansen CL, Stevens-Lapsley JE. Incorporating Specific Functional Strength Integration Techniques to Improve Functional Performance for Veterans After Total Hip Arthroplasty: Protocol for a Randomized Clinical Trial. Phys Ther. 2019 Nov 25;99(11):1453-1460. doi: 10.1093/ptj/pzz109. PMID 31392991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from orthopedic clinics.
Period: Overall Study
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Started | 45 | 50
Completed | 41 | 45
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON) | Total
Number analyzed (Participants) | 45 | 50 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.2) | 64.5 (7.0) | 63.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants declined to provide their sex.
  Participants
    number analyzed (Participants) | 45 | 48 | 93
    Female | 15 | 34 | 49
    Male | 30 | 14 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 41 | 40 | 81
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 50 | 95
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — units: kg/m2
  kg/m^2 | 28.9 (4.8) | 27.7 (4.2) | 28.3 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test (6MW)
Description: Patients will perform a 6MW test, which assesses how far a patient walks in 6 minutes. The 6MW test was chosen as the primary outcome because it captures performance over a period of time that best mimics community ambulation with activities of daily living. Higher numbers indicate better function. The 6MW test is reliable and valid in the post-THA population and can detect small changes in function after THA. 6MW will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in 6MW from baseline to intervention end-point (after 8 week intervention; POST2)
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 41 | 45
meters | 252.4 [194.2 to 310.5] | 207.0 [151.5 to 262.5]

2. Secondary Outcome: 4 Meter Walk (4MW)
Description: The 4MW test measures the time to walk 4 meters and has been used to generate gait speed values, which have been associated with morbidity and mortality in older adults. Higher numbers indicate better speed values. Participants will perform the 4MW with instructions to walk in their "normal, everyday pace." 4MW will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in 4MW from baseline to intervention end-point (after 8 week intervention; POST2)
Population: The number analyzed for this outcome measure differs from the overall number analyzed due to some participants not meeting ability/safety criteria at assessment timepoint.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 40 | 45
seconds | -0.69 [-0.83 to -0.56] | -0.54 [-0.67 to -0.41]

3. Secondary Outcome: 30 Second Sit-to-stand (30 STS)
Description: The 30 second sit-to-stand test assesses functional lower extremity strength and endurance, and has been validated and found reliable in older adults at various physical activity levels and physical independence levels. Higher numbers indicate better lower extremity strength and endurance. 30 STS will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in 30 STS from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of sit to stand cycles
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 37 | 41
number of sit to stand cycles | 4.22 [3.07 to 5.36] | 3.39 [2.30 to 4.47]

4. Secondary Outcome: Functional Gait Assessment (FGA)
Description: Participants will also perform the FGA, which is a 10-item objective outcome measure designed to measure dynamic balance while walking in the presence of external demands, and will provide information on patients' stability before and after THA. The FGA has been shown to be a reliable and valid measure, effective in classifying fall risk in older adults and predicting unexplained falls. Scores range from 0-30, with higher scores indicating better functions. FGA will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in FGA from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 39 | 45
score on a scale | 3.71 [2.66 to 4.76] | 3.63 [2.65 to 4.61]

5. Secondary Outcome: Isometric Strength
Description: Isometric strength of the quadriceps and hip abductor muscles will be assessed on a handheld dynamometer. All strength testing will be performed in positions that minimize the risk of hip dislocation post-operatively, while still allowing for optimal trunk and pelvic stabilization. Isometric quadriceps strength testing will be performed in sitting at 0 hip flexion and 60 knee flexion. Isometric hip abduction strength testing will be performed in side lying at 0 flexion/extension and 0 hip abduction. Testing will include warm-up repetitions, followed by three separate maximal voluntary isometric contractions while receiving visual and verbal feedback. Strength will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in strength from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: kg force/kg body mass
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 39 | 45
kg force/kg body mass
  Involved Hip Abductor: number analyzed (Participants) | 38 | 45
  Involved Hip Abductor | 0.15 [0.02 to 0.28] | 0.06 [-0.07 to 0.18]
  Uninvolved Hip Abductor: number analyzed (Participants) | 39 | 44
  Uninvolved Hip Abductor | 0.14 [0.04 to 0.24] | 0.02 [-0.07 to 0.11]
  Involved Quad Strength | 0.64 [0.43 to 0.86] | 0.54 [0.34 to 0.75]
  Uninvolved Quad Strength | 0.31 [0.09 to 0.53] | 0.23 [0.03 to 0.44]
  Involved Hamstring: number analyzed (Participants) | 39 | 41
  Involved Hamstring | 0.24 [0.14 to 0.34] | 0.18 [0.08 to 0.28]
  Uninvolved Hamstring: number analyzed (Participants) | 39 | 42
  Uninvolved Hamstring | 0.09 [-0.01 to 0.20] | 0.06 [-0.04 to 0.16]

6. Secondary Outcome: Modified Trendelenburg Test
Description: Patients will complete hip abductor endurance testing using a static single-limb balance test,. This modified Trendelenburg test assesses neuromuscular control during single limb stance and indicates the ability of the lateral hip muscles to maintain pelvic control during closed-chain, functional tasks and therefore serves as a measure of hip abductor muscle endurance. This test will be performed using a high-speed motion-capture system to assess lateral pelvic tilt. Differences in length of time pelvic control is maintained will be analyzed from preoperative to postoperative assessments during the single-limb task on the surgical leg. Trendelenburg will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in Trendelenburg test from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 38 | 45
seconds | 4.27 [2.09 to 6.46] | 2.81 [0.80 to 4.81]

7. Secondary Outcome: Peak Internal Hip Abduction Moment
Description: Surgical limb peak internal hip abduction moment will be calculated with 3-D instrumented motion analysis. Continuous internal hip abduction moments will be calculated during functional task performance using a standard inverse dynamics approach integrating kinematic and kinetic data using Visual 3D software (C-Motion, Germantown, MD). Peak internal hip moment during activity is a measurement of muscle activity during the task and provides insight to how muscles are activated during the task. Since the intervention exercise program targeted improving recruitment of the hip abductor moments during gait and other functional tasks, we calculated internal hip abduction moments. From the continuous hip moments, peak surgical limb internal hip abduction moments during the Loading Response phase of the stance period of the walking trials will be collected. Moments will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in moment from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: kg force/kg body mass
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 39 | 44
kg force/kg body mass
  Involved Hip Abduction Moment | 3.44 [1.04 to 5.84] | 0.62 [-1.62 to 2.85]
  Uninvolved Hip Abduction Moment | 3.27 [1.23 to 5.30] | 0.42 [-1.50 to 2.32]

8. Secondary Outcome: ActiGraph
Description: ActiGraph activity monitors assess physical activity (PA) using accelerometry, which allows objective evaluation of the relative volume (steps/day) and intensity (activity counts) of physical activity with high validity and reliability. Each participant will wear the ActiGraph for at least 4 days at all time points to assess average daily PA (steps/day). Higher number of steps indicates higher level of physical activity. PA will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in physical activity from baseline to intervention end-point (after 8 week intervention; POST2)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 23 | 25
steps per day | 892 [152 to 1631] | 1014 [306 to 1722]

9. Secondary Outcome: Veterans RAND 12-item Health Survey (VR-12)
Description: The Veterans RAND (VR-12) is a reliable, self-report survey for assessing health-related quality of life. The questions in this survey correspond to seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS) which then provides an important contrast between the respondents' physical and psychological health status. Each component score is summarized from 0 to 100, with a higher score indicating a better outcome. VR-12 scores will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in VR-12 from baseline to intervention end-point (after 8 week intervention; POST2)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 41 | 45
score on a scale
  Physical Component Score | 15.2 [12.7 to 17.7] | 16.4 [14.0 to 18.8]
  Mental Component Score | 4.16 [2.02 to 6.30] | 3.82 [1.78 to 5.86]

10. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The WOMAC is a self-report questionnaire that assesses the impact of osteoarthritis on pain, stiffness, and disability. The WOMAC has been shown to be a valid, reliable, and responsive instrument often used in clinical trials. Scores range from 0-96, with higher scores indicating more pain, stiffness, and disability. WOMAC scores will also be assessed at mid-intervention (POST1, 4 weeks) and 26-week evaluation (POST3).
Time Frame: Change in WOMAC from baseline to intervention end-point (after 8 week intervention; POST2)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 41 | 45
score on a scale | -35.0 [-39.2 to 30.9] | -38.4 [-42.4 to -34.5]

11. Secondary Outcome: Patient Activation Measure (PAM)
Description: The PAM survey assesses patient knowledge, skill, and confidence for self-management, as self-efficacy exhibits a positive relationship with preventive actions and health outcomes. The Continuous Score is a composite score of the available 10 items, ranging from 0-100, wherein a higher score indicates a higher activation (better outcomes). The PAM Level is the mean of the 4 Categorical Levels, wherein a higher score indicates a higher activation (better outcomes). Categorical Level 1: disengaged and overwhelmed; Categorical Level 2: becoming aware but still struggling; Categorical Level 3: taking action & gaining control; Categorical Level 4: maintaining behaviors & pushing further. Specific cut offs for each Categorical Level are unavailable, as scoring is proprietary.
Time Frame: Assessed at baseline only
Population: Two participants chose not to complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 44 | 49
score on a scale
  Continuous | 71.3 (12.7) | 70.6 (14.2)
  PAM Level | 3.34 (0.57) | 3.27 (0.70)

12. Secondary Outcome: Patient Activation Measure (PAM) Categorical
Description: The PAM survey assesses patient knowledge, skill, and confidence for self-management, as self-efficacy exhibits a positive relationship with preventive actions and health outcomes. The Categorical Levels are frequency distribution of the scores between 1-100, wherein a higher Categorical Level indicates a higher activation (better outcomes). Categorical Level 2: becoming aware but still struggling; Categorical Level 3: taking action & gaining control; Categorical Level 4: maintaining behaviors & pushing further. Specific cut offs for each Categorical Level are unavailable, as the scoring is proprietary.
Time Frame: Assessed at baseline only
Population: Two participants chose not to complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 44 | 49
Participants
  Categorical Level 2 | 2 | 7
  Categorical Level 3 | 25 | 22
  Categorical Level 4 | 17 | 20

13. Secondary Outcome: Motivation Scale
Description: The motivation scales asks the participant "How motivated do you feel to participate in physical therapy?", and rating on a 0 (not at all motivated) to 10 (very motivated) scale. Higher scores indicate higher level of motivation.
Time Frame: Quantification at Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 45 | 50
score on a scale | 9.42 (1.4) | 9.28 (1.1)

14. Other Pre Specified Outcome: Pain Levels at Rest and With Activity
Description: Patients will report pain levels at rest and with activity (numerical pain rating scale [NPRS; 0= no pain, 10= worst possible pain]) at all testing timepoints.
Time Frame: Quantification at baseline, POST1 (after 4 weeks intervention), POST2 (after 8 weeks intervention), and POST3 (26 weeks after initiating rehabilitation)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 45 | 50
score on a scale
  Involved Limb Pain at Rest Baseline | 4.4 (2.368352) | 4.62 (2.406539)
  Uninvolved Limb Pain at Rest Baseline | 1.022222 (1.936361) | 0.7 (1.328648)
  Involved Limb Pain with Activity Baseline | 4.822222 (2.405381) | 4.64 (2.472378)
  Uninvolved Limb Pain with Activity Baseline | 0.711111 (1.791675) | 0.1 (0.416497)
  Involved Limb Pain at Rest Post1: number analyzed (Participants) | 37 | 42
  Involved Limb Pain at Rest Post1 | 1.297297 (1.596261) | 0.952381 (1.305754)
  Uninvolved Limb Pain at Rest Post1: number analyzed (Participants) | 37 | 42
  Uninvolved Limb Pain at Rest Post1 | 0.756757 (1.816673) | 0.047619 (0.308607)
  Involved Limb Pain with Activity Post1: number analyzed (Participants) | 37 | 42
  Involved Limb Pain with Activity Post1 | 1.108108 (1.760426) | 0.904762 (1.393531)
  Uninvolved Limb Pain with Activity Post1: number analyzed (Participants) | 37 | 42
  Uninvolved Limb Pain with Activity Post1 | 08.10811 (1.853493) | 0.095238 (0.484367)
  Involved Limb Pain at Rest Post2: number analyzed (Participants) | 41 | 45
  Involved Limb Pain at Rest Post2 | 0.902439 (1.462957) | 0.533333 (0.990867)
  Uninvolved Limb Pain at Rest Post2: number analyzed (Participants) | 41 | 45
  Uninvolved Limb Pain at Rest Post2 | 0.780488 (2.07981) | 0.133333 (0.547723)
  Involved Limb Pain with Activity Post2: number analyzed (Participants) | 41 | 45
  Involved Limb Pain with Activity Post2 | 0.707317 (1.346178) | 0.555556 (1.139289)
  Uninvolved Limb with Activity Pain Post2: number analyzed (Participants) | 41 | 45
  Uninvolved Limb with Activity Pain Post2 | 0.804878 (2.170478) | 0.044444 (0.208409)
  Involved Limb Pain at Rest Post3: number analyzed (Participants) | 31 | 35
  Involved Limb Pain at Rest Post3 | 1.096774 (1.325515) | 0.200000 (0.531369)
  Uninvolved Limb Pain at Rest Post3: number analyzed (Participants) | 31 | 35
  Uninvolved Limb Pain at Rest Post3 | 0.806452 (1.621097) | 0.171429 (0.513678)
  Involved Limb with Activity Pain Post3: number analyzed (Participants) | 31 | 35
  Involved Limb with Activity Pain Post3 | 0.580645 (1.176837) | 0.285714 (0.621735)
  Uninvolved Limb Pain with Activity Post3: number analyzed (Participants) | 31 | 35
  Uninvolved Limb Pain with Activity Post3 | 0.451613 (1.206613) | 0.114286 (0.529785)

15. Other Pre Specified Outcome: Injury
Description: Patient report musculoskeletal injury history at all testing timepoints.
Time Frame: POST1 (after 4 weeks intervention), POST2 (after 8 weeks intervention), and POST3 (26 weeks after initiating rehabilitation)
Population: The number analyzed for this outcome measure differs from the overall number analyzed due to some participants not completing the assessment timepoint.
Measure: Number; unit: participants
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 41 | 45
participants
  Injury Post1: number analyzed (Participants) | 37 | 42
  Injury Post1 | 3 | 5
  Injury Post2 | 0 | 5
  Injury Post3: number analyzed (Participants) | 31 | 35
  Injury Post3 | 5 | 2

16. Other Pre Specified Outcome: Falls
Description: Patients will report falls at all testing timepoints.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: falls
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
Number analyzed (Participants) | 45 | 50
falls
  Falls Post1: number analyzed (Participants) | 37 | 42
  Falls Post1 | 0.108108 (0.3148) | 0.119048 (0.395239)
  Falls Post2: number analyzed (Participants) | 41 | 45
  Falls Post2 | 0.02439 (0.156174) | 0.088889 (0.358166)
  Falls Post3: number analyzed (Participants) | 33 | 37
  Falls Post3 | 0.225806 (0.61694) | 0.257143 (0.741337)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Functional Strength Integration (FSI) | Control Group (CON)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/50
Other Adverse Events (participants affected / at risk) | 3/45 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Strength Integration (FSI) (N=45) | Control Group (CON) (N=50)
Falls (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02920866/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02920866/ICF_001.pdf